CLINICAL TRIAL: NCT03840668
Title: Healthy Living Through Personalized Monitoring of Eyelid Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: Ngee Ann Polytechnic Singapore (Unknown)
Responsible Party: Principal Investigator, Louis Tong, Clinician-Scientist, Senior Consultant, Singapore National Eye Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R1507/6/2018; 2018/2102 (Registry Identifier: SingHealth CIRB)
Record Dates: First submitted 2018-12-03; First posted 2019-02-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Dry Eye
Keywords: USB eyemask
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dry eye (Experimental): Participants who will be using the USB-powered eye mask.
  Interventions: Device: USB Eye Mask

INTERVENTIONS:
Device: USB Eye Mask — To evaluate the acceptance of the USB eye mask via questionnaire and also to monitor the use of USB eye mask over a period of 2 months.

SUMMARY:
Portable USB-powered eyemasks provide convenience to dry eye sufferers to perform eyelid warming at home. Such eyemasks can be plugged into a copyrighted device developed in collaboration with Ngee Ann Polytechnic that tracks patients' usage. This revolutionary device transmits a signal and is sent to a cloud system whenever the device is used and activity of usage will be recorded. The cloud database only allows access to administrator and will be password protected. You or your physician can monitor the frequency of eyelid warming over a long period.

DETAILED DESCRIPTION:
Dry eye is a very common condition that can cause blurring of vision associated with reading, grittiness, eyelid heaviness and poor tolerance of light. Up to 80% of dry eye is due to blocked oil glands in the eyelids known as Meibomian Gland Dysfunction (MGD) and scientific studies have shown that sustained eyelid warming at 40-42°C for at least 8 minutes a day is effective to control this condition and increase the tear film layer thickness.

Portable USB-powered eyemasks provide convenience to dry eye sufferers to perform eyelid warming at home. Such eyemasks can be plugged into a copyrighted device developed in collaboration with Ngee Ann Polytechnic that tracks patients' usage. This revolutionary device transmits a signal and is sent to a cloud system whenever the device is used and activity of usage will be recorded. The cloud database only allows access to administrator and will be password protected. You or your physician can monitor the frequency of eyelid warming over a long period. To further encourage eyelid warming to be performed more frequently, the signal can also be sent to a participating games server which hastens progress in the game. Thus, addiction to online games, which usually worsens symptoms of dry eye can now be a way to treat dry eye.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 21 years or older.
2. Subject must have severe MGD
3. Subject must be willing to answer the questions in the questionnaire
4. Subject must be willing to use the USB-powered eyemask as instructed
5. Subject must have the ability to provide informed consent
6. Subject must be willing to come back for follow-up visit

Exclusion Criteria:

1. Any other specified reason as determined by the clinical investigator.
2. Is pregnant, lactating or planning a pregnancy.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Acceptance of USB eyemask questionnaire | 2 months +/-14 days
  Participants will be asked to answer some questionnaires on acceptance and evaluation of USB eye mask

CONTACTS AND LOCATIONS:
Overall Officials: Louis Tong, PhD, Principal Investigator — Singapore Eye Research Institute
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore